CLINICAL TRIAL: NCT05819723
Title: Analgesia Produced by Erector Spinae Block and Incidence of Postoperative Delirium After Hip Fracture Surgeries
Brief Title: Erector Spinae Block and Incidence of Postoperative Delirium After Hip Fracture Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Associate professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MS 99/2023
Record Dates: First submitted 2023-03-29; First posted 2023-04-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Delirium in Old Age

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- spinal anesthesia only (Active Comparator): The spinal anaesthesia will be done under a complete aseptic technique induced using 3ml bupivacaine 0.5% with 25μg fentanyl
  Interventions: Other: CAM score
- spinal anesthesia with erector spinae block (Active Comparator): The spinal anaesthesia will be done under a complete aseptic technique induced using 3ml bupivacaine 0.5% with 25μg fentanyl, then erector spinae block will be given The transverse process of the 4th lumbar vertebra will be identified 4-6 cm laterally to the midline. An echogenic needle will be inserted using the out-of-plane technique until it touches the transverse process. Following negative aspira¬tion, 20 ml of 0.25% bupivacaine will be injected
  Interventions: Other: CAM score

INTERVENTIONS:
Other: CAM score — The CAM scores assess the presence of delirium rapidly and accurately and also differentiates delirium from other cognitive impairment with a sensitivity of 94-100% and specificity of 90-95%.
  It is an algorithm that consists of four features:
  (i) Acute and fluctuating variation in mental status, (ii) Inattention, (iii) Incoherent or disorganized thinking, and (iv) Altered level of consciousness. CAM scores indicate delirium if the first two features are present and either the third or fourth feature is present.

SUMMARY:
Postoperative pain is a significant risk factor for delirium. This clinical trial will search whether analgesia produced by erector spinae block in elderly patients undergoing hip fracture surgeries reduces delirium or not!

DETAILED DESCRIPTION:
This randomized controlled trial will include 120 elderly patients American Society of Anesthesiologists physical status I-II, aged more than 60 years old and undergoing fracture hip surgeries.

all patients will be examined for preoperative cognitive impairment using the short form of the Confusion Assessment Method Survey (CAM) and the long form will be used postoperatively.

The CAM scores is an algorithm that consists of four features:

(i) Acute and fluctuating variation in mental status, (ii) Inattention, (iii) Incoherent or disorganized thinking, and (iv) Altered level of consciousness.CAM scores indicate delirium if the first two features are present and either the third or fourth feature is present.

Patients with a delirium of CAM score>1 will be excluded from the study. also, patients will be asked to rate their baseline pain levels using the numeric rating scales (NRS) from "no pain" to "worst possible pain". patients will be randomly divided into two equal groups Group 1: spinal anaesthesia only. Group 2: spinal anaesthesia with erector spinae block. In both groups, basic monitoring in the form of non-invasive blood pressure (NIBP), pulse oxygen saturation (SPO2)and 5-lead electrocardiogram (ECG) will be attached in the operating room(OR)

The spinal anaesthesia will be done in both groups under a complete aseptic technique induced using 3ml bupivacaine 0.5% with 25μg fentanyl.

At the end of the operation patients in group 2 will receive the block at the lateral position.

The transverse process of the 4th lumbar vertebra will be identified 4-6 cm laterally to the midline. An echogenic needle will be inserted using the out-of-plane technique until it touches the transverse process. Following negative aspiration, 20 ml of 0.25% bupivacaine will be injected.

patients will be monitored in the PACU for at least one hour by NIBP, SPO2, and ECG and any abnormality will be recorded and managed accordingly.

The cognitive functions will be re-evaluated one hour after the recovery from the surgery in PACU using the CAM scores. and on the first and the second days postoperatively using CAM score for occurrence and severity of cognitive dysfunction if present. Then every symptom will be rated and listed in the CAM-S as absent (0, mild (1), or severe (2), where higher scores indicate more severe delirium and patients with POD will be followed up and managed properly by neurologists. Patients in the two groups will be compared regarding the incidence and severity of delirium on the first and second postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years.
* American Society of Anesthesiologists physical status I, II.
* Patients undergoing hip fracture surgeries under spinal anaesthesia

Exclusion Criteria: • History of neurological or psychiatric disease.

* Allergy to local anaesthetics.
* Infection in the injection area.
* Regular medication with tranquillizers and/or antidepressants.
* CAM scores II-VI.
* Delayed fracture surgeries more than 48 hours.
* Intraoperative blood loss of more than 1000 ml.
* Patient refusal.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
post operative delirium | first days postoperative
  occurrence and severity of cognitive dysfunction

SECONDARY OUTCOMES:
complications from erector spinae block | on the first and the second days postoperative
  block failure, haematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt